CLINICAL TRIAL: NCT00719342
Title: Effect of Breathing a Mixture of 92% O2 + 8% CO2 on Flicker Induced Blood Flow Changes in Ocular Perfusion
Brief Title: Effect of Breathing a Mixture of 92% Oxygen (O2) + 8% Carbon Dioxide (CO2) on Flicker Induced Blood Flow Changes in Ocular Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-030606
Record Dates: First submitted 2008-07-01; First posted 2008-07-21 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Flicker-induced Vasodilatation
Keywords: Retinal vessel diameter; Flicker-induced vasodilatation; Optic nerve head blood flow; Ocular Physiology; Regional Blood Flow
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Oxygen + Carbondioxide — Mixture of 92 % oxygen and 8 % carbon dioxide for inhalation
  Other Names: O² + CO²; Oxymix
Other: full field flickering light at 12.5 Hz — 1 minute stimulation with full field flickering light at 12.5 Hz during measurement of vessel diameters and measurement of blood flow.

SUMMARY:
It has been shown that diffuse luminance flicker increases retinal and optic nerve head blood flow. This indicates that a neuro-vascular coupling between neural activity and blood flow exists in the retina as described previously for the brain. Although a lot of mediators such as NO, pO2, pCO2, H+ and K+ have been proposed, the mechanism of this coupling is still a matter of controversy. However, it has been shown in an animal experiment, that an increase in blood flow, evoked by diffuse luminance flicker stimulation is paralleled by decrease in pO2 in the tissue. In a recently performed study we could show that breathing of 100% O2 did not influence flicker induced changes in the retina and optic nerve head. However, breathing of 100% oxygen also leads to a pronounced vasoconstriction of the retinal vessels and in turn to a increased tension of the vessel wall. Recent evidence indicates that a combination of 92% O2 and 8% CO2 can, at least partially, counteract the vasoconstrictory effect of O2 and increases tissue pO2. Thus, in this study the investigators set out to investigate the flicker light induced increase in blood flow under a mixture of O2/CO2 .

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow | 1 hour
Retinal vessel diameters | 1 hour

SECONDARY OUTCOMES:
blood pressure | 1 hour
pulse rate | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria